CLINICAL TRIAL: NCT02969174
Title: Clinical Professor of Shanghai Tongji Hospital
Brief Title: Establish a Non-invasive Prenatal Genotyping and Extraction Technology to Diagnose and Treat the HDN.
Status: Approved for marketing | Type: Expanded Access
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Liming Cheng, The President of Shanghai Tongji Hospital, Shanghai Tongji Hospital, Tongji University School of Medicine
Other Study IDs: ShangjiTongjiHsxk
Record Dates: First submitted 2016-11-03; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: HDFN

INTERVENTIONS:
Other: zimin Lu,Guo Sa — chengzhong Liu

SUMMARY:
To establish a genotyping and extraction technology of non invasive prenatal diagnosis for fetal blood group genotype from cell-free fetal DNA in peripheral blood of pregnant women.

To achieve prenatal accurate identification of fetal blood group genotypes，and provide credible theoretical evidence for the prenatal diagnosis and treatment of hemolytic disease of newborn (HDN).

DETAILED DESCRIPTION:
Establish a Non-invasive Prenatal Genotyping and Extraction Technology to Diagnose and Treat the HDN.

ELIGIBILITY:
Inclusion Criteria:

blood samples of pregnant couples,gender/nation/region is unlimited.

Exclusion Criteria:

adipose or hemolytic samples,overdue samples,unidentified samples

Ages: 12 Weeks to 38 Weeks | Sex: All
Age Groups: Child